CLINICAL TRIAL: NCT06941766
Title: Efficacy and Safety of Iparomlimab and Tuvonralimab (QL1706) in the Treatment of Intermediate Trophoblastic Tumors: A Prospective, Multicenter, Single-arm Trial
Brief Title: Iparomlimab and Tuvonralimab (QL1706) for Intermediate Trophoblastic Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Shengjing Hospital (Other); Obstetrics & Gynecology Hospital of Fudan University (Shanghai Red House Ob & Gyn Hospital) (Unknown); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Henan Cancer Hospital (Other Government); Gansu Provincial Maternal and Child Health Care Hospital (Other); Dalian women and children's medical group (Unknown); The First Affiliated Hospital of Xiamen University (Other); Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, xiang yang, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITT01
Record Dates: First submitted 2025-04-15; First posted 2025-04-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Intermediate Trophoblastic Tumor
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- QL1706±chemo (Experimental): Cohort A: QL1706: 5 mg/kg, intravenous (IV) infusion, every 3 weeks (Q3W), administered on Day 1 (D1).Chemotherapy Options: FAEV, EMA/EP, EMA/CO, or TP/TE.
  Cohort B: QL1706: 5 mg/kg, IV infusion, Q3W (D1).
  Interventions: Drug: QL1706; Drug: Chemotherapy

INTERVENTIONS:
Drug: QL1706 — 5 mg/kg, IV infusion, Q3W (D1)
Drug: Chemotherapy — FAEV, EMA/EP, EMA/CO, or TP/TE.

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of Iparomlimab and Tuvonralimab (QL1706), a dual-targeting immunotherapy (anti-PD-1/CTLA-4), in patients with intermediate trophoblastic tumors (ITT).

The main questions it aims to answer are:

Does QL1706 improve complete response (CR) rates (primary endpoint) and survival outcomes? What are the safety profiles of QL1706 in ITT, including immune-related adverse events? Participants will receive QL1706 (5 mg/kg IV, Q3W) ± chemotherapy (FAEV/EMA/EP/EMA/CO/TP-TE). They will also receive Maintenance therapy post-hCG normalization. Efficacy is assessed via serial β-hCG tests, imaging (every 9-12 weeks), and biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

Females aged 18-70 years. Histologically confirmed placental site trophoblastic tumor (PSTT) or epitheloid trophoblastic tumor (ETT)

For Cohort A:

Stage IV disease (treatment-naïve）, recurrent, or chemotherapy-resistant disease

For Cohort B:

Stage I-III disease requiring adjuvant chemotherapy post-biopsy/surgery, meeting ≥1 of: Abnormal β-hCG 2 weeks post-surgery; Incomplete resection; High-risk features includes: Interval from last pregnancy ≥48 months; Deep myometrial invasion; Mitotic count >5/HPF; Tumor necrosis.

ECOG score 0-1. Signed informed consent.

Organ Function Requirements:

Hematologic:

WBC ≥3.0×10⁹/L ANC ≥1.5×10⁹/L Platelets ≥80×10⁹/L Hemoglobin ≥8.0 g/dL Creatinine ≤1.5×ULN Total bilirubin ≤1.5×ULN (or direct bilirubin ≤ULN if total bilirubin >1.5×ULN) AST/ALT ≤2.5×ULN INR/PT/aPTT ≤1.5×ULN (or within therapeutic range if on anticoagulants).

Exclusion Criteria:

Life expectancy <3 months. Non-gestational trophoblastic tumors. Active malignancy (except if cured ≥3 years prior). Prior immune checkpoint therapy (anti-PD-1/L1, CTLA-4, ICOS, CD40, etc.) or cell-based immunotherapies.

Active autoimmune disease requiring systemic treatment (past 2 years). Exceptions: Hormone replacement (e.g., thyroxine), physiologic corticosteroids (≤10 mg/day prednisone equivalent).

Active inflammatory bowel disease (e.g., Crohn's, ulcerative colitis). Systemic corticosteroids (>10 mg/day prednisone equivalent) within 14 days. Allowed: Topical/inhaled steroids, prophylactic steroids for contrast allergy.

HIV/AIDS.

Active hepatitis:

HBV DNA >1,000 IU/mL (unless on stable antiviral therapy with DNA <1,000 IU/mL).

HCV RNA-positive (unless cured). Active tuberculosis (screening required if suspected). Uncontrolled severe infection (e.g., sepsis, pneumonia requiring hospitalization).

Cardiovascular disease: NYHA Class III/IV heart failure or LVEF <50%. Uncontrolled hypertension (≥140/90 mmHg despite treatment). Unstable angina, myocardial ischemia, or arterial thromboembolism (≤6 months).

Interstitial lung disease (history or active). Malabsorption syndromes (e.g., chronic diarrhea, bowel obstruction) or GI perforation/fistula (≤6 months).

Psychiatric/social conditions impairing consent or compliance. Allogeneic transplant history. Live vaccines ≤30 days prior to QL1706 or planned during study. Hypersensitivity to monoclonal antibodies or protocol-specified chemotherapies. Pregnancy/lactation. Other conditions deemed to compromise patient safety or study integrity.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — ITT only occurs in women
Enrollment: 20 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-04-16 (Estimated); Study Completion 2028-04-16 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate | up to one year
  Percentage of patients achieving CR, as defined by normalization of serum hCG (≤5 IU/L for ≥4 weeks)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to one year
  Proportion of evaluable patients achieving CR + Partial Response (PR) (serum hCG decline >50% from baseline but without normalization)
Disease Control Rate (DCR) | up to one year
  Proportion of evaluable patients with CR + PR + Stable Disease (SD) (serum hCG fluctuation ≤50% from baseline)
Rate of Progression-Free Survival (PFS) | up to one year
  Time from treatment initiation to radiographic progression (RECIST v1.1) or death from any cause
Rate of Overall Survival (OS) | up to one year
  Time from first dose to death from any cause
Concentration of anti-Müllerian hormone (AMH) to assess ovarian function | up to one year
  Ovarian function as assessed by anti-Müllerian hormone (AMH)
Number of Participants with treatment-related Adverse Events [Safety and Tolerability] | up to one year
  Determine frequency and severity of adverse events as assessed by NCI CTCAE (Version 5.0)
Quality of life of cancer patients by questionnaire | up to one year
  Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30(EORTC QLQ-C30) It consists of 30 questions across multiple scales, including a global health status scale and functional scales (physical, role, emotional, cognitive, and social functioning) to evaluate daily activities and well-being. Symptom scales cover common issues like fatigue, pain, and nausea. The tool's reliability and validity make it effective for measuring the impact of cancer and its treatments, with additional disease-specific modules available for tailored assessments.
Cancer specific rehabilitation by questionnaire | up to one year
  Assessed by Cancer rehabilitation evaluation system-short form (CARES-SF) It is a brief, validated questionnaire designed to assess emotional well-being, functional status, and social support in cancer survivors. It is specifically tailored to evaluate the psychosocial and functional adjustment of individuals after cancer treatment, focusing on areas such as emotional distress, social functioning, and physical well-being. The tool is often used in oncology and rehabilitation settings to monitor the quality of life and recovery of cancer patients during and after treatment. It is concise, easy to administer, and provides valuable insights into the holistic needs of cancer survivors.
Reproductive concerns after cancer by scale | up to one year
  Assessed by Reproductive Concerns After Cancer (RCAC) scale. The minimum and maximum values are 18 and 90 respectively, and a higher score means a higher level of reproductive concern or anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No